CLINICAL TRIAL: NCT07262047
Title: Characterization and Health Related Quality of Life Among Children With Inborn Error of Immunity
Brief Title: Quality of Life Among Children With Inborn Error of Immunity
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ali, doctor, Sohag University
Other Study IDs: Soh-Med-25-9-14MS
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of Life Assessment — Administration of standardized quality-of-life questionnaires (e.g., PedsQL) to children with primary immunodeficiency and/or their caregivers.

SUMMARY:
In this study, we aim to assess the QOL of pediatric IEI patients compared with healthy controls and to determine different factors affecting QOL in these patients.

DETAILED DESCRIPTION:
Inborn Errors of Immunity (IEI) are a group of approximately 430 heterogeneous immunity disorders that are characterized by decreased immunity at the innate level involving disorders of phagocytosis and the complement system or at the adaptive level including B-cell, T-cell, or combined immunodeficiencies [1]. Another updated phenotypic classification of IEI suggested by the International Union of Immunological Societies (IUIS) in 2021, identifies 10 categories that include immunodeficiencies affecting cellular and humoral immunity (severe combined immunodeficiency: SCID or combined immunodeficiency), combined immunodeficiencies with associated or syndromic features (such as congenital thrombocytopenia, DNA repair defects, etc.), predominantly antibody deficiencies with recurrent bacterial infections (IgG, IgA, IgM deficiencies), diseases of immune dysregulation and autoinflammatory disorders [2]. The most common of these are the primary antibody deficiencies [3] which include common variable immunodeficiency, IgA, or IgG deficiency, X-linked agammaglobulinemia and other specific antibody deficiencies [1].

Severity of IEI also vary between asymptomatic as in the case of IgA deficiencies to life-threatening forms such as SCID (sever combined immunodeficiencies) [4]. Diagnosed IEI patients are more susceptible to acquiring infections, malignancies, autoimmunity, and lympho-proliferative disorders [5]. Most IEI are diagnosed at an early age but can present later in adulthood. Early detection and management are associated with better outcomes. Hence, screening [6-8] and employing a high level of suspicion is a key factor in improving detection rates of IEI [9]. Newborn screening for treatable and severe forms of IEI is now a common practice in many countries. As for management, the mainstay of treatment for most antibody deficiency is regular intravenous or subcutaneous immunoglobulin therapy [10-11] and bone marrow transplantation for combined immunodeficiencies; these therapies are associated with an improved quality of life (QOL) [12-13].

The burden imposed by IEI on patients is huge and encompasses both physical and emotional consequences especially due to the severity and chronicity of the disorder. Children with IEI have lower health related quality of life (HRQOL) scores [14], and more limitations in physical and social functioning [15-18]. The literature also shows a high disease burden for IEI which includes a higher number of hospitalizations per year, emergency room visits, monthly visits to clinics as well as family monthly expenses related to the disease and absenteeism from school or work [19]. The most widely used tool for assessing HRQOL in pediatric IEI patients is the Pediatric Quality of Life Inventory (PedsQL) which measures 4 domains, which are physical, emotional, social, and school functioning as reported by either parent or child [20]. Several studies assess the QOL of pediatric IEI patients and reveal a poor quality of life that is associated with delayed diagnosis and type of disease. There is a paucity of literature on the QOL of pediatric IEI patients, even though it is more common in upper Egypt where consanguinity is a prevalent occurrence. Therefore, this study is the first to assess the QOL of pediatric IEI patients using the PedsQL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* children from 6 years untill 18 years

Exclusion Criteria:

* failed to get a consent not appropriate age

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children diagnosed with primary immunodeficiency who are followed at participating immunology clinics or hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Arabic version of PedsQL, version 4 | At enrollment
  The tool is composed of 23 items that cover the following domains: physical, emotional, social, and school functioning. Each item is on a 5-point Likert scale ranging between 0 and 4 (0= never, 1= almost never, 2= sometimes, 3= often, 4= almost always). Scores are linearly transformed to a 0- to 100- point scale (4 = 0, 3 = 25, 2 = 50, 1 = 75, 0= 100) and higher scores reflect a better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: eman mohamed fahmy, Study Director — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bousfiha A, Jeddane L, Al-Herz W, Ailal F, Casanova JL, Chatila T, Conley ME, Cunningham-Rundles C, Etzioni A, Franco JL, Gaspar HB, Holland SM, Klein C, Nonoyama S, Ochs HD, Oksenhendler E, Picard C, Puck JM, Sullivan KE, Tang ML. The 2015 IUIS Phenotypic Classification for Primary Immunodeficiencies. J Clin Immunol. 2015 Nov;35(8):727-38. doi: 10.1007/s10875-015-0198-5. Epub 2015 Oct 7. PMID 26445875
- [Background] de Vries E, Driessen G. Educational paper: Primary immunodeficiencies in children: a diagnostic challenge. Eur J Pediatr. 2011 Feb;170(2):169-77. doi: 10.1007/s00431-010-1358-5. Epub 2010 Dec 18. PMID 21170549
- [Background] Tangye SG, Al-Herz W, Bousfiha A, Cunningham-Rundles C, Franco JL, Holland SM, Klein C, Morio T, Oksenhendler E, Picard C, Puel A, Puck J, Seppanen MRJ, Somech R, Su HC, Sullivan KE, Torgerson TR, Meyts I. Human Inborn Errors of Immunity: 2022 Update on the Classification from the International Union of Immunological Societies Expert Committee. J Clin Immunol. 2022 Oct;42(7):1473-1507. doi: 10.1007/s10875-022-01289-3. Epub 2022 Jun 24. PMID 35748970
- [Background] Picard C, Al-Herz W, Bousfiha A, Casanova JL, Chatila T, Conley ME, Cunningham-Rundles C, Etzioni A, Holland SM, Klein C, Nonoyama S, Ochs HD, Oksenhendler E, Puck JM, Sullivan KE, Tang ML, Franco JL, Gaspar HB. Primary Immunodeficiency Diseases: an Update on the Classification from the International Union of Immunological Societies Expert Committee for Primary Immunodeficiency 2015. J Clin Immunol. 2015 Nov;35(8):696-726. doi: 10.1007/s10875-015-0201-1. Epub 2015 Oct 19. PMID 26482257